CLINICAL TRIAL: NCT02817295
Title: Bariatric Surgeries in Elderly
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of Surgery department, Assuta Medical Center
Other Study IDs: 2015073
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- elderly: patients underwent bariatric surgery and are above 65 years old
  Interventions: Other: clinical measurements
- non-elderly: patients underwent bariatric surgery and are below 65 years old
  Interventions: Other: clinical measurements

INTERVENTIONS:
Other: clinical measurements — follow up on the number of complications, revisions, hospitalization and co-morbidities

SUMMARY:
an examination of the different aspects of bariatric surgery in elderly in comparison with non-elderly patients.

DETAILED DESCRIPTION:
the study examines the success rate, complications, revisions, days of hospitalization and co-morbidities in elderly and in non-elderly patients that underwent bariatric surgery in our medical center

ELIGIBILITY:
Inclusion Criteria:

bariatric surgery

Exclusion Criteria:

below 18 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwent baritaric surgery
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of complications. | six months
  data collection and analysis will be ended in six months. data will be collected from the medical records.
Number of revisions | six months
  data collection and analysis will be ended in six months. data will be collected from the medical records.
Number of days of hospitalization | six months
  data collection and analysis will be ended in six months. data will be collected from the medical records.
Incidence of co-morbidities | six months
  data collection and analysis will be ended in six months. data will be collected from the medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No